CLINICAL TRIAL: NCT03422302
Title: Measuring the Effectiveness of a Continuous Positive Airway Pressure (CPAP) Device to Reduce Tumor Motion and Increase Lung Volume Expansion in Patients Undergoing Stereotactic Body Radiotherapy (SBRT) for Tumors That Move With Respiration
Brief Title: Continuous Positive Airway Pressure Device or Deep Inspiration Breath Hold in Reducing Tumor Motion in Patients Undergoing Stereotactic Body Radiation Therapy for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1105; NCI-2018-00884 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1105 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Lung Carcinoma; Malignant Respiratory Tract Neoplasm; Metastatic Malignant Neoplasm in the Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Continuous Positive Airway Pressure; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (CT simulation, CPAP, DIBH, SBRT, BiPAP) (Experimental): Patients undergo free-breathing, DIBH, and CPAP CT simulation scans. If patient has difficulty exhaling on CPAP, then patient undergo BiPAP CT simulation. The attending physician then compares all 3 simulation treatment plans (free-breathing, DIBH, and CPAP/BiPAP) and determines which method to use during SBRT. If CPAP/BiPAP is chosen as preferred method, patients wear CPAP/BiPAP over 1 hour prior to SBRT, then again during SBRT over 30-60 minutes. All other patients complete free-breathing or DIBH during SBRT over 30-60 minutes.
  Interventions: Device: Biphasic Positive Airway Pressure; Procedure: Computed Tomography; Procedure: Continuous Positive Airway Pressure; Procedure: Deep Inspiration Breath Hold; Radiation: Radiation Therapy Treatment Planning and Simulation; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Device: Biphasic Positive Airway Pressure — Receive BiPAP
  Other Names: BiPAP; Biphasic positive airway pressure (BiPAP)
Procedure: Computed Tomography — Undergo CT simulation scans
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Continuous Positive Airway Pressure — Receive CPAP
  Other Names: Continuous positive airway pressure (CPAP); CPAP
Procedure: Deep Inspiration Breath Hold — Complete DIBH
  Other Names: DIBH
Radiation: Radiation Therapy Treatment Planning and Simulation — Undergo CT simulation scans
  Other Names: Radiation Therapy Treatment Planning/Simulation
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This pilot phase I/II trial studies how well a continuous positive airway pressure device or deep inspiration breath hold works in reducing tumor movement in patients undergoing stereotactic body radiation therapy (SBRT) for lung cancer. The continuous positive airway pressure device works by blowing air into the lungs while patients wear a face mask or nozzle to help expand their airways and lungs. Deep inspiration breath hold is a standard technique that uses active breath-holding to restrict movement of the body. Using a continuous positive airway pressure device may work better than deep inspiration breath hold in lowering the amount of tumor movement during stereotactic radiation body therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the two methods of tumor motion management, continuous positive airway pressure (CPAP) and deep inspiration breath hold (DIBH) and to estimate the decrease in tumor motion from free breathing for CPAP and DIBH.

SECONDARY OBJECTIVES:

I. To determine if CPAP is a more time-efficient option for tumor motion management than is DIBH.

Ia. Determine if CPAP is better tolerated by patients than is DIBH. Ib. Determine the reproducibility of lung expansion and tumor motion reduction by CPAP.

Ic. Determine if the dosimetric coverage of the tumor and the sparing of the normal tissues with CPAP is comparable to that with DIBH.

Id. Measure treatment time differences between CPAP and breath hold (DIBH) treatments.

OUTLINE:

Patients undergo free-breathing, DIBH, and CPAP CT simulation scans. If patient has difficulty exhaling on CPAP, then patient undergo biphasic positive airway pressure (BiPAP) CT simulation. The attending physician then compares all 3 simulation treatment plans (free-breathing, DIBH, and CPAP/BiPAP) and determines which method to use during SBRT. If CPAP/BiPAP is chosen as preferred method, patients wear CPAP/BiPAP over 1 hour prior to SBRT, then again during SBRT over 30-60 minutes. All other patients complete free-breathing or DIBH during SBRT over 30-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The patient will receive stereotactic body radiotherapy in the Thoracic Radiation Oncolcogy Service at MD Anderson.

Exclusion Criteria:

* The patient has a contra-indication for using a CPAP device.
* The patient has not signed a study-specific informed consent for this study.
* The patient is uncooperative.
* The patient has reduced consciousness.
* The patient has sustained trauma or burns to the face.
* The patient has undergone any facial, esophageal, gastric or sinus surgery within the last 3 months.
* The patient has idiopathic pulmonary fibrosis (IPF) as documented in their medical history.
* Adults who are unable to consent, individuals who are not yet adults, pregnant women and prisoners will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of decrease in tumor motion | Up to 10 days
  Paired t-test will be used to compare continuous positive airway pressure (CPAP) to deep inspiration breath hold (DIBH) in the decrease of tumor motion from free breathing. Linear regression may be used to evaluate the difference between CPAP and DIBH in the decrease of tumor motion from free breathing with the adjustment of important demographic and clinical variables in the model.

SECONDARY OUTCOMES:
Increase in lung volume | Up to 10 days
  Increase in lung volume to be determined by using DIBH or CPAP from free breathing. Linear regression may be used to evaluate the difference between CPAP and DIBH in the increase of lung volume from free breathing with the adjustment of important demographic and clinical variables in the model. The study will summarize the data with mean, standard deviation, median and range for continuous variables, and frequency count and percentage for categorical variables
Assessment of time to deliver the planned radiation dose by using the most appropriate method | Up to 10 days
  The study will summarize the data with mean, standard deviation, median and range for continuous variables, and frequency count and percentage for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Julianne M Pollard, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org